CLINICAL TRIAL: NCT05000541
Title: Observation of the Effects of Guideline-driven Lifestyle Interventions, Including Use of a Red-yeast Based Nutraceutical , in Subjects With Hypercholesterolemia at Low-moderate Cardiovascular Risk Not Requiring a Drug Therapy
Brief Title: Observation of the Effects of Guideline-driven Lifestyle Interventions, Including Use of a Red-yeast Based Nutraceutical
Status: Completed | Type: Observational
Sponsor: Mylan Inc. (Industry)
Collaborators: Mylan Österreich GmbH (Unknown); Mylan Germany GmbH (Unknown); Mylan Healthcare Sp. z o.o. (Unknown)
Responsible Party: Sponsor
Organization: Viatris Inc. (Industry)
Other Study IDs: 3319
Record Dates: First submitted 2021-08-04; First posted 2021-08-11 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-04

CONDITIONS: Hypercholesterolemia
MeSH Terms: conditions — Hypercholesterolemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Armolipid-L/Armolipid Plus-L: Armolipid-L used for participants in Germany and Poland Armolipid Plus-L used for participants in Austria

SUMMARY:
The objective of the present multinational, multicentre, prospective, scientific study is to confirm that prescription of a low-dose red yeast-based nutraceutical.

DETAILED DESCRIPTION:
The objective of the present multinational, multicentre, prospective, scientific study is to confirm that prescription of a low-dose red yeast-based nutraceutical significantly increases the LDL-C lowering effect of guideline-driven lifestyle interventions in subjects with hypercholesterolemia at low-moderate cardiovascular risk not requiring a drug therapy.

ELIGIBILITY:
Inclusion Criteria:

* Age between 25 and 75 years;
* In primary prevention for low-moderate CV risk, with diet and physical exercise to control raised LDL-C level, for at least 3 months;
* LDL-C > 100 mg/dL (2.6 mmol/L), < 190 mg/dL (4.9 mmol/L)
* CV risk SCORE <5% (based on SCORE chart according to figure I for Poland respective figure 2 for Austria and Germany in the ESC/EAS guideline 2019);
* Triglyceride <400 mg/dL;
* Advised to use nutraceutical as part of the lifestyle intervention as per guideline and within the product label (i.e. posology as in product label);
* Written informed consent.

Exclusion Criteria:

* Subjects being treated or who have been treated for up to 3 months before the start of the study with lipid-lowering drugs or nutraceuticals including functional foods for which lipid-lowering effects are known (e.g. fish oil, sterol-containing yoghurts etc.);
* Subjects involved in other clinical studies with pharmaceutical products
* Known laboratory evidence of either liver, muscle, thyroid or kidney dysfunction;
* Subjects with prior history of cardiovascular events or with high cardiovascular risk equivalents;
* Uncontrolled hypertension (systolic blood pressure >190 mmHg or diastolic blood pressure >100 mmHg);
* Pregnancy and breastfeeding.

Ages: 25 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects to be enrolled are subjects already in primary prevention for CVD for raised LDL-C and who, according to the intervention strategies recommended in Table 5 of the ESC/EAS guidelines (lifestyle interventions, consider drug if uncontrolled) had been prescribed, in the previous 3 months, only dietary advices and physical exercise.
Sampling Method: Non-Probability Sample
Enrollment: 259 (Actual)
Dates: Start 2020-12-08 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2023-10-31 (Actual)

PRIMARY OUTCOMES:
Mean change from baseline in LDL-C | 3 months
  Mean change from baseline in LDL-C at 3 months

SECONDARY OUTCOMES:
Subjects' adherence to the prescribed lifestyle interventions measured on Visual Analogue Scale (VAS) | at 3 months and 6 months
  Subjects' adherence (at 3 months and 6 months) to the prescribed lifestyle interventions measured on Visual Analogue Scale (VAS); minimum 0mm, maximum 100mm; higher value means better adherence

CONTACTS AND LOCATIONS:
Locations (7):
- Austria (2):
  - Ordination, Unterhautzenthal
  - Ordination, Vienna
- Germany (5):
  - Medical Practice, Bexbach
  - Medical Practice, Deggingen
  - Medical Practice, Frankfurt
  - Medical Practice, Görlitz
  - AmBeNet GmbH, Leipzig